CLINICAL TRIAL: NCT04158921
Title: Control:Diabetes - a Mobile App to Improve Glycemic Control in Patients With Diabetes
Brief Title: Control:Diabetes Pilot Study I
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Alexander Turchin, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: controldiabetes01
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Insulin Treated Type 2 Diabetes Mellitus; Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus; Insulin Therapy; Glycemic Control; Hyperglycemia; Hypoglycemia; Health Education; Self-Management; Lifestyle
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Hyperglycemia; Hypoglycemia; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The Control:Diabetes mobile app for Diabetes self-management. (Other): This is a single arm open label pilot clinical trial that will assess patient-reported blood glucose levels before and after using the Control:Diabetes mobile app.
  Interventions: Other: Control:Diabetes mobile app

INTERVENTIONS:
Other: Control:Diabetes mobile app — The Control:Diabetes app will encourage patients to: a) predict their blood glucose level at a particular time point in the future (e.g. the next morning); then b) enter their actual blood glucose levels when that time (the next morning) comes; and c) enter reasons for the discrepancy between prediction and reality, if the prediction was significantly (e.g. > 20%) different from the actual measurement. We hypothesize that by repeatedly encouraging disassembly of blood glucose changes into individual reasons (cognitive task analysis) while providing an incentive in the form of being able to more accurately predict blood glucose levels (operant conditioning), the app will prompt the patient to learn how various internal and environmental factors affect their blood glucose. They will then be able to adjust their behavior and medications to improve their blood glucose control.

SUMMARY:
This is a single arm open label pilot clinical trial that will assess patient-reported blood glucose levels before and after using the Control:Diabetes mobile app, while collecting user feedback and recommendations for further improvements to the app functionality and user interface. This study will enroll approximately 70 individuals with insulin-treated diabetes mellitus. The study will include two online surveys (baseline and exit), one study initiation phone call, and will also collect data entered by the users into the mobile app.

DETAILED DESCRIPTION:
The objectives of this study are to:

* Test the hypothesis that patients with diabetes mellitus treated with insulin and elevated blood glucose will achieve better glycemic control after using the Control:Diabetes mobile app.
* Test the hypothesis that patients with diabetes mellitus treated with insulin and frequent hypoglycemia will achieve lower frequency of hypoglycemia after using the Control:Diabetes mobile app.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of Type 1 Diabetes or Type 2 Diabetes
* Treatment with multiple daily insulin injections (MDII) or continuous subcutaneous insulin infusion (CSII)
* Baseline HbA1c between 7% and 10.5% (as reported by the participant) and/or self- reported frequency of symptomatic hypoglycemia ≥ 3 times / week
* Ownership of a smartphone running either Android or iOS operating system with an active data plan

Exclusion Criteria:

* Using a closed loop insulin delivery system (Medtronic 670G or OpenAPS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
The mean change in blood glucose. | Measured between the first two weeks and the last two weeks of the study.
  As recorded by the patient in the app.

SECONDARY OUTCOMES:
The change in the number of hypoglycemic episodes. | Measured every week between the two weeks prior to the study entry and the last two weeks of study follow-up.
  Number of low blood sugar episodes as reported in the study surveys.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No